CLINICAL TRIAL: NCT02453828
Title: The Effects of Implementing an Anesthesia Information Management System Guided Intraoperative Anesthesia Care Transition Checklist on Postoperative Complications: A Randomized Trial
Brief Title: Intraoperative Anesthesia Care Transition Checklist
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has requested for this study be closed due to technical issues
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15-192
Record Dates: First submitted 2015-03-09; First posted 2015-05-27 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Checklist (Experimental): after non-cardiac surgery, patients will have current standard-of-care anesthesia handover during anesthesia transitions in care with an additional, electronically pre-populated checklist displayed on the anesthesia record keeping system
  Interventions: Procedure: Non-cardiac surgery
- Standard of Care (Active Comparator): after non-cardiac surgery, patients will have current standard-of-care anesthesia handover during anesthesia transitions in care
  Interventions: Procedure: Non-cardiac surgery

INTERVENTIONS:
Procedure: Non-cardiac surgery — patients having non-cardiac surgery

SUMMARY:
Perioperative management decisions must often be made quickly and rely on practitioners having relevant facts at hand. During transitions of patient care between anesthesia providers, known as "handovers," information may not be completely or faithfully communicated, consequently impairing the provider's ability to intervene correctly in response to subsequent events. Checklists have consistently proven to be effective at enhancing communications during handovers, but whether anesthesia checklists improve patient outcomes has yet to be proven. The investigators propose to randomize intraoperative anesthesia provider handovers to standard practice (no specific format) or to a handover checklist presented by a decision-support system in conjunction with the investigators electronic record. Specifically, the investigators will test the hypothesis that incorporating a largely pre-populated handover checklist into transitions of intraoperative anesthesia care decreases a composite of mortality and serious cardiovascular, respiratory, gastrointestinal, urinary, and infectious complications.

DETAILED DESCRIPTION:
The modern team-based approached to patient care often involves transitioning care between providers. Critical details may be lost during transition, or handovers, resulting in delays, inefficiencies, suboptimal care, or even patient harm. The Joint Commission on Hospital Accreditation declared that communication failures are the root cause of almost two-thirds of all sentinel events. The World Health Organization similarly listed "communication during patient care handover" as one of the highest patient safety initiatives. The consequence of ineffectual communication may be especially detrimental during surgery when patients are often unstable and post-handover decisions must be made quickly and accurately. In a preliminary study the investigators observed an 8% increase in odds of experiencing major in-hospital morbidity or mortality per for each intraoperative handover.

Checklists have been used for transitions of care in a variety of areas; orthopedic trauma, urological robotic surgeries, and emergency departments. The field of anesthesia has also embraced the use of checklists, especially in the handover to intensive care units. Post-anesthesia checklists have been the particular focus of anesthesia providers in recent years. Post-operative checklists clearly enhance information transfer, but have only been evaluated using historical controls which do not account for bias. The anesthesia area most lacking valid studies is intraoperative handovers.

Anesthesia-specific intraoperative handovers differ because the interaction is primarily between anesthesia providers while surgery continues without disruption. To date, there has only been one proposed checklist for intraoperative handovers between anesthesia providers and it has not been prospectively evaluated. A randomized study with contemporaneous controls, utilizing an anesthesia specific, electronically pre-populated checklist measuring objective "hard" outcomes will address the limitations of previous studies.

The investigators propose to test the hypothesis that incorporating an electronic handover checklist during transitions of intraoperative anesthesia care reduces serious complications. Specifically, the investigators will quantify the effect of a handover checklist on adverse outcomes as defined by a composite of mortality and serious cardiovascular, respiratory, gastrointestinal, urinary, and infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* non-cardiac surgery

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7348 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
a composite of in-hospital mortality and 6 major morbidities including serious cardiac, respiratory, gastrointestinal, urinary, bleeding, and infectious complications | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Leif Saager, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States